CLINICAL TRIAL: NCT06245655
Title: A Randomized Controlled Trial of Transcutaneous Electrical Nerve Stimulation (TENS) for Treatment of IUD Insertion Pain
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) for IUD Insertion Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Lauren Kus, Complex Family Planning Fellow, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-23-01562; SFP17-UL4 (Other Grant/Funding Number: Society of Family Planning)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TENS (Active Comparator): For the Active TENS group, the device will be set to 80 Hz (hfTENS) and device intensity (0-8) will be titrated to patient comfort, as is the standard protocol for TENS use.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Placebo TENS (Placebo Comparator): For the placebo TENS group, setup will be identical, but the device will not be turned on.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — TENS 7000 digital TENS unit, a low cost, over the counter, battery operated device with high consumer ratings. The handheld device works by transmitting an electronically generated topical stimulus to a specified area on the body to alter response to pain signals and promote endogenous endorphin release for pain reduction.

SUMMARY:
This study is a double-blind, randomized, placebo-controlled trial to evaluate the use of high frequency TENS for pain control during IUD insertion. Transcutaneous electrical nerve stimulation (TENS) is a relatively low-cost, low-risk, non-pharmacologic intervention for pain management. Previous studies have found that TENS reduces pain associated with other outpatient gynecological procedures. Participants will be randomized in a 1:1 ratio to either active treatment or placebo (placebo TENS) and record pain scores using a 100 mm visual analog scale (VAS) at the time of IUD insertion. The same device will be used for both active and placebo treatment.

DETAILED DESCRIPTION:
The researchers will recruit eligible participants from patients who opt for IUD initiation during ambulatory care visits to the Mount Sinai Complex Family Planning service at Mount Sinai Hospital, Mount Sinai Beth Israel, Mount Sinai Morningside, and Mount Sinai West. Allocation to treatment will be based on a 1:1 blocked randomization scheme stratified by parity. A member of the research/clinical team other than the person performing IUD insertion will identify the treatment allocation assigned to the corresponding subject ID. The team member will set up the TENS unit accordingly by applying pads to the participant and initiating treatment with the correct settings. When setup is complete (<5 minutes), the person performing the IUD insertion and other clinical staff assisting with the procedure will enter the exam room with no knowledge of TENS treatment assignment to insert the IUD.

REDCap, a HIPAA-compliant, secure web application used for building and managing online surveys and databases, will be used for data collection in this study. Participants will complete electronic surveys in REDCap during the study. The first survey is a baseline survey to collect demographics as well as medical, obstetric, and gynecologic history and other characteristics prior to the IUD insertion procedure.

IUD insertion will be performed by complex family planning faculty and fellows, as well as OB/GYN residents on their family planning rotation. A research staff member will be within reach of the study participant during the procedure to collect pain scores using a visual analog scale (VAS) presented on an iPad.

The second survey will have a visual analog scale for study participants to rate their pain between 0 and 100 at the following timepoints during IUD insertion:

1. Baseline
2. Immediately after bimanual exam
3. Immediately after speculum insertion
4. Immediately after tenaculum placement
5. Immediately after uterine sounding
6. Immediately after IUD insertion
7. 5 minutes after speculum removal

The third survey will ask participants about reflections on their experience with IUD insertion and acceptability of the TENS device. Participation in the study is expected to only last one day, the day of IUD insertion.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in the study, an individual must meet all the following criteria:

* Presenting for IUD initiation during ambulatory care visits to the Mount Sinai Complex Family Planning service
* Provision of signed and dated informed consent form for IUD Insertion
* English speaking and age 18 or older
* Opting for either LNG 52mg or copper T380A IUD
* Stated willingness to comply with all study procedures

Exclusion Criteria:

* Contraindication to IUD initiation (i.e. pregnancy, current pelvic infection, distorted uterine anatomy)
* Contraindication or allergy to ibuprofen
* History of a chronic pain disorder
* Recent opioid use in the previous 30 days
* History of a cardiac arrhythmia
* History of heart disease (i.e. atrial fibrillation, congestive heart failure)
* Presence of an implantable device with an electrical discharge (i.e. pacemaker)
* BMI > 50 (class IV obesity)
* History of TENS use
* Planned pain intervention outside standard of care (i.e. paracervical block) OR pre-procedure use of non-standard pain medication (i.e. benzodiazepines, muscle relaxers, gabapentin, benadryl)
* History of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analog Scale | Day 1 (Day of IUD Insertion)
  Pain Visual Analog Scale - full scale from 0-100, higher score indicates higher level of pain

SECONDARY OUTCOMES:
Post Procedure Survey | Day 1 (Day of IUD Insertion)
  Factors other than exposure to TENS associated with higher reported pain, Acceptability of the TENS device. Questions answered as yes or no. This is not a scale and has no min or max score.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Kus, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - Center for Women's Health and Midwifery, New Haven, Connecticut
  - Yale Family Planning Clinic, New Haven, Connecticut
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No
Individual participant data meta-analysis for this study will not be done. De-identified individual participant data will be analyzed according to the statistical plan mentioned in the study protocol for manuscript preparation and journal publication. Individual participant data will be shared within the study team. Also, IPD will be shared with the IRB according to institutional guidelines.

DOCUMENTS (1):
  • Informed Consent Form (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT06245655/ICF_000.pdf